CLINICAL TRIAL: NCT06157307
Title: A Pilot Study Comparing the Efficacy of Four Different Methods of Performing External Aortic Compression in Healthy Women After Caesarean Section
Brief Title: Four Different Methods of Performing External Aortic Compression After Caesarean Section
Acronym: KEXAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Annette Aronsson, Doctor, Region Stockholm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: AAronsson
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Postpartum Hemorrhage
Keywords: Aortic compression
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test subjects (Experimental): Four different hand placements for aortic compression.
  Interventions: Device: Aortic compression

INTERVENTIONS:
Device: Aortic compression — Aortic compression with four different methods on each participants

SUMMARY:
After childbirth, bleeding from the uterus occurs, which can quickly become very profuse if the uterus does not contract. Annually, around 80000 women die because profuse bleeding associated with childbirth, mainly in low -and middle income countries. By pressing a fist on the outside of the abdomen in the umbilical plane (aortic compression) the abdominal artery is compressed, which directly reduces the bleeding from the uterus and any bleeding from the birth canal.

The goal of this small clinical trial is to compare four different ways of performing aortic compression in healthy women directly after a planned uncomplicated cesarean section.

The main questions aim to answer are:

* Is there a difference in how well aortic compression works, defined as cessation of blood flow in the inguinal artery measured by ultrasound, when applying aortic compression with the fist positioned in the transverse plane or longitudinally, compared to the fingertips and a fist protector
* Does the researcher experience a difference between the four different methods? The study takes place in the operating room immediately the cesarean sectio is complete. The participant will then still have the effect of the spinal anesthetic. The researcher begin the trial by recording vital signs: heart rate and electrical activity, blood pressure and the amount of oxygen in the blood. Ultrasound will be used to see the blood flow in the right inguinal artery. If everything is normal, the researcher will apply aortic compression in four different ways.

The researcher will start aortic compression with the fingertips, then with a fist placed lengthwise. After that with the fist across the abdomen and then with a fist protector. At each occasion there will be a maximum of 5 seconds of total occlusion of the abdominal artery. Cessation of blood flow in the inguina artery becomes the criterion for total compression of the abdominal artery below the umbilicus. After the trial, the participant will be transferred to the post-operative ward, where, in addition to standard monitoring, you are also observed for 30 minutes by of the researcher.

The study is carried out at Karolinska University Hospital and takes approximately 20 minutes, including preparation.

There are no clinical benefits for the participants. Increased knowledge of different ways of performing aortic compression can contribute to better treatment of women with profuse bleeding after childbirth.

DETAILED DESCRIPTION:
This is a pilot study comparing the efficacy of four different methods of performing external aortic compression in healthy women after caesarean section. In patients with severe postpartum hemorrhage (PPH) external compression of the abdominal aorta, may temporize the bleeding and thus reduce morbidity and mortality. PPH is a serious obstetric emergency and the single most important cause of maternal mortality globally The most common causes of PPH are uterine atony followed by placental disorders, retained placenta and membranes, birth trauma and coagulation defects. The World Health Organization defines PPH as the blood loss of ≥500 mL within the first 24 hours after delivery. Severe PPH is defined ≥1000 mL. The majority of PPH occur within 4 hours. The incidence of severe PPH is reported to vary between 1 - 5% of all births, depending upon the diagnostic criteria applied. Early diagnosis and management are critical in preventing maternal deaths. Manual external aortic compression is a technique that can be applied immediately to reduce bleeding from the uterus or birth canal by reducing its blood supply as aorta is compressed against the column through the abdominal wall.

Objectives and hypotheses of the clinical investigation In this pilot study the primary objective is cessation of femoral artery blood flow when applying external aortic compression in women immediately after they have given birth by caesarean section with the fingertips, the fist placed longitudinally, with the fist placed transversally compared with the padded fist protector At each of the four methods of compressing aorta, the cessation of the flow in the femoral artery and hemodynamic parameters will be registered. The primary endpoint is the cessation of pulsation in the femoral artery measured by ultrasound. Reduction of the femoral artery blood flow can be assumed to be a surrogate marker for the reduction of blood flow in the aorta and thus to areas below the compressed aorta.

Secondary objective is to evaluate if there a difference in the investigator experience between the four different methods. The ExAC fist protector has been developed to facilitate the manual external aortic compression used to temporarily reduce or stop postpartum bleeding. The fist protector provides a soft padding of the fist that allows any unevenness to be reduced when aorta is compressed between the boney surface of fist and the spinal column and facilitates herby a complete compression. The fist protector will be put on the fist of the researcher who will apply external aortic compression. The researcher will otherwise do the maneuver as usual.The investigator will evaluate if the fist protector makes it easier to perform the maneuver. The participant will evaluate if the fist protector leads to less discomfort

In this pilot study the main research questions are as follows:

Is there a difference in the efficacy, defined as cessation of blood flow in the femoral artery measured by ultrasound doppler, when applying external aortic compression with the fingertips, the fist placed longitudinally, with the fist placed transversally Sample size calculation and justification Six healthy, female participants will be included in the study. There has been no sample size calculation. This is a small pilot study, and the device is to be modified prior to further investigation.

PERFORMANCE AND SAFETY VARIABLES:

The heart rate (HR) and cardiac rhythm, blood pressure (BP) and oxygen saturation will be registered, and the femoral artery identified at the level just below the inguinal ligament using the ultrasound scanning. The sequence of aortic compression at the level of umbilicus will be applied for maximum 5 seconds of complete occlusion in the following manner:

1. Performed with the fingertips.
2. Performed with with the fist placed longitudinally.
3. Performed with the fist placed transversally.
4. Performed with ExAC compression fist protector At each of the four methods of compressing aorta the flow in the femoral artery and hemodynamic parameters will be registered Anticipated adverse device effects External aortic compression is associated with pain and discomfort. To reduce the discomfort for the participants it is an advantage that the participant has a spinal anesthesia. For this study we have chosen to include women after c-section when they still have a spinal anesthesia.

Anticipated adverse events of the investigations include:

* Discomfort/pain.
* Slightly increase in blood pressure induced by aortic compression. Six healthy women who have undergone uncomplicated caesarean sections are selected as subjects because the discomfort and inconvenience for these women will be less prominent compared to recently vaginally delivered women. Immediately after the operation has been completed, the women remain on the operating table in the right position and it is easy carry out the study. Participants Inclusion criteria

  * Normal pregnancy
  * No ongoing medication
  * Age 18 - 35
  * BMI 18.5-30
  * Proficient Swedish language skills
  * Uncomplicated caesarean sectio Exclusion criteria
  * Tobacco/Nicotine use
  * Any ongoing medication
  * Any chronic disease except seasonal allergy
  * Previous abdominal surgery
  * Complicated caesarean section The researcher team consists of 3 people. A principal investigator and two researchers from Karolinska University Hospital Solna.

One researcher will perform the aortic compression, one will evaluate the flow in the femoral artery using ultrasound scanning. The third researcher will help the principal investigator to obtain the measurements.

Recruitment and screening The parturient will be recruited among patients who have a planned caesarean section at Karolinska University Hospital Solna. The patient will get verbal and written information about the study and will have the opportunity to ask questions. After the participant has agreed to participate, she will be asked to sign and date an informed consent. Enrolled to the study will be after the caesarean sectio. Preparation of subject and continuous safety monitoring of subject The infant can stay on the mothers chest after the caesarean section and this will be preferred. By the mothers request the baby will be taken care of by the father or the midwife.

Following measurements will be monitored during the investigation:

* Pulse-oximeter
* Non-invasive blood pressure (NIBP)
* Electrocardiogram (ECG)
* Heart rate
* Flow in the femoral artery Baseline measurements The investigator registers heart rate (HR) and cardiac rhythm, blood pressure (BP) and oxygen saturation. The coinvestigator will identify the femoral artery at the level just below the inguinal ligament using the ultrasound scanning. The ultrasound sequences will be recorded for each individual and stored. Experimental measurements Once the baseline measurements are complete, the participant will rest for 2 minutes before the actual experiment commences. The sequence of aortic compression will be applied in the following manner for maximum 5 seconds of complete occlusion. The compressions will be done at the level of umbilicus.

  1. Performed with the fingertips.
  2. Minimum 2 minutes of no occlusion.
  3. Performed with the fist placed longitudinally.
  4. Minimum 2 minutes of no occlusion.
  5. Performed with the fist placed transversally.
  6. Minimum 2 minutes of no occlusion.
  7. Performed with ExAC compression fist protector Variables that will be registered

  <!-- -->

  1. Baseline measurements

     1. Pulse-oximeter
     2. Non-invasive blood pressure (NIBP)
     3. Electrocardiograph (ECG)
     4. Heart rate In case of failure to compress the aorta by closed fist or ExAC fist protector a maximum of three new attempts with repositioning will be done. A failure of occlusion of the aorta will be registered. Baseline measurements (blood pressure, heart rate, and oxygen saturation) will be re-registered between the three experimental maneuvers. This will ensure correct baseline measurements for each maneuver. Follow up After the study, the subjects will be observed for 30 minutes. All subjects will be informed to contact the primary investigator (mobile phone number provided) in case of any concerns related to the investigation for the first 7 days. Data Collection The clinical investigation data will be collected on paper CRF completed by one of the researchers Participant Records and Source Data The data will be recorded directly in the CRF, which will then be considered as source data. The origin of source data in the investigation will be further specified in a separate document . It is the responsibility of the investigation site to record essential information in the medical records in accordance with national regulations and requirements:
* Study code
* Participant ID code
* That informed consent for participating in the study was obtained
* All visits during the investigation period
* All adverse events (AE)/adverse device events (ADE)s
* Treatments and medications The Investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data recorded.

ELIGIBILITY:
Inclusion Criteria:

* Normal pregnancy
* No ongoing medication
* BMI 18.5-30
* Proficient Swedish language skills
* Uncomplicated caesarean sectio

Exclusion Criteria:

* Tobacco/Nicotine use
* Any ongoing medication
* Any chronic disease except seasonal allergy
* Previous abdominal surgery
* Complicated caesarean section

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-08 (Estimated)

PRIMARY OUTCOMES:
Femoral blood flow | 60 seconds
  The primary endpoint is the cessation of pulsation in the femoral artery measured by ultrasound.

SECONDARY OUTCOMES:
investigator experience | 60 seconds
  a difference in the investigator experience between the four different methods

CONTACTS AND LOCATIONS:
Overall Officials: Annette Aronsson, MD,PhD, Principal Investigator — Karolinska University Hospital

IPD SHARING:
Plan to Share IPD: No